CLINICAL TRIAL: NCT07316855
Title: Safety and Efficacy of Bioresorbable Iron-Based Covered Stent System for the Treatment of Coarctation of the Aorta: A Single-Center Clinical Study
Brief Title: Evaluating the Feasibility of Bioresorbable Iron-Based Covered Stent: A Clinical Trial
Acronym: CoA-ICS-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shubo Song (Other)
Collaborators: Central China Fuwai Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor-Investigator, Shubo Song, Associate Chief Physician, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CoA-ICS-I; 251111314300 (Other Grant/Funding Number: The Key Research and Development Project of Henan Province, China)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coarctation of the Aorta
Keywords: Coarctation of the Aorta; Bioresorbable; covered stent; Biodegradable; iron-based
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Intervention Model Description: single-center, single-group, target value, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TBSI-CoA (Experimental): Transcatheter bioresorbable iron-based covered stent implantation for the patients with coarctation of the aorta
  Interventions: Device: Implantation of Bioresorbable Iron-based Covered Aortic Stent

INTERVENTIONS:
Device: Implantation of Bioresorbable Iron-based Covered Aortic Stent — A novel bioresorbable iron-based covered stent for coarctation of the aorta

SUMMARY:
A single-center, feasible clinical study to Evaluate the Treatment of Iron Bioresorbable Covered Scaffold System in patients with Coarctation of the Aorta Diseases

DETAILED DESCRIPTION:
There is a feasibility study. Ten subjects are intended to participate in this study and without control group. The Iron Bioresorbable Covered Scaffold System will be implanted surgically. Follow-up will be conducted at 1 month, 3 months, 6 months and 12 months post-procedure. The primary endpoint is the rate of no restenosis of the stent at 12 months post-procedure [Defined on a per target lesion basis]

ELIGIBILITY:
Inclusion Criteria:

1. Patient must between 1 and 60 years old

   Patients being clinically diagnosed with CoA or patients with post-operative anastomotic stenosis after CoA surgery，meanwhile meeting one of the following conditions:

   A：Pressure gradient of Carctation in a calm state. B：The degree of aortic stenosis is not less than 50% (degree of Carctation Of the Arota = (diameter of adjacent normal segment of blood vessel - residual vessel lumen diameter of stenotic segment)
   * diameter of adjacent normal segment of blood vessel×100% ) C：Peak velocity of echocardiographic Doppler in the CoA≥2.5m/s
2. The patients and their families have high compliance, sign the informed consent and willing to undergo 1-year follow-ups and related examinations.
3. The patient's expected lifespan is more than one year after successful treatment with the stent.
4. Reference vessel (diameter of the adjacent normal segment vessel ) diameter：4-16mm

Exclusion Criteria:

1. Patients with a history of iron overload or iron disorder, such as hereditary hemochromatosis, etc.
2. Patients with cardiopulmonary function that cannot tolerate surgery, such as severe heart failure (NYHA Grade III and above) that cannot be controlled by active medical treatment.
3. Patients with known allergy to contrast agent, iron and its degradation products.
4. Patients with hemorrhagic disorders
5. Patients with contraindications on antiplatelet agents and anticoagulant therapy.
6. Patients with thrombosis at the vascular wall of target lesion and the distal or proximal location of the lesion.
7. Patients with known severe renal or hepatic insufficiency, which are unsuitable for index procedure
8. Target lesion to be treated where stent was implanted previously.
9. Patients with severe stenosis or excessive tortuosity in the targeted vessel, or anatomical abnormalities, which predict the device will have difficulty reaching the target lesion.
10. Other conditions that are unfavorable for stent delivery or balloon expansion.
11. Patient who have already participated in another clinical trial, and have not yet completed or withdrawn within 3 months before the screening period of this trial.
12. Patients who are not suitable for participating the trial as per investigator judgement.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1.Rate of no stent restenosis[Defined on a per target lesion basis] | at 12 months post-procedure
  Definition of stent restenosis: If the pressure difference within the stent on transthoracic echocardiography is 50% higher than the result of transthoracic echocardiography at 0-1 days post-procedure, will be considered as suspected restenosis.
2.Acute Procedure Success | after the stent is delivered to the target lesion site and expanded during the procedure
  Definition of Acute Procedure Success：Meeting any one of the following standards after the stent is delivered to the target lesion site and expanded during the procedure A.The pressure difference between the proximal and distal ends of the stenosis decreased by≥50% ,detected by right heart catheterization after the stent being placed.
  B.The inner diameter of the original stenotic segment of the blood vessel increases by ≥50% after the stent is placed，detected by pulmonary artery angiography after the stent being placed.

SECONDARY OUTCOMES:
1.Acute Technical Success | after the stent is delivered to the target lesion site and expanded during the procedure
  Technical Success
2.Rate of no stent restenosis | at 1,3, 6 months post-index procedure
  defined on a per target lesion basis，no stent restenosis
3.The rate of device related Major Adverse Events ( MAE ) and Serious Adverse Events（SAE） | at 1,3, 6, 12months post-index procedure
  device related Major Adverse Events ( MAE ) and Serious Adverse Events（SAE）
4.The rate of unexpected secondary surgical or interventional procedures | at 1,3, 6, 12months post-index procedure
  unexpected secondary surgical or interventional procedures (excluding the expected secondary intervention procedures)
5.Rate of Stent Thrombosis | at 1,3, 6, 12months post-index procedure
  Stent Thrombosis
6.Rate of all-cause mortality | at 1,3, 6, 12months post-index procedure
  all-cause mortality
7.The rate of displacement after stent implantation | at 1,3, 6, 12months post-index procedure
  displacement after stent implantation
8.The rate of Major Adverse Events ( MAE ) and Serious Adverse Events（SAE）during the study | at 1,3, 6, 12months post-index procedure
  Major Adverse Events ( MAE ) and Serious Adverse Events（SAE）during the study

CONTACTS AND LOCATIONS:
Overall Officials: Taibing Fan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
The patient's age, weight, as well as the ultrasound and CT data during the perioperative period and follow-up period can be shared, but the patient's name, hospital number and ID number and other confidential information cannot be shared.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: The International Committee of Medical Journal Editors can access the IPD